CLINICAL TRIAL: NCT03247283
Title: Pharmacokinetics and Metabolism of [14C] BMS-986205 in Healthy Male Participants
Brief Title: Pharmacokinetics and Metabolism Study in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CA017-052A
Record Dates: First submitted 2017-08-07; First posted 2017-08-11 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — linrodostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Oral Dose of BMS-986205 (Experimental)
  Interventions: Drug: BMS-986205

INTERVENTIONS:
Drug: BMS-986205 — Carbon 14 tagged BMS-986205

SUMMARY:
Phase 1 Phamacokinetic and metabolism study of BMS-986205 in healthy males

ELIGIBILITY:
Inclusion Criteria:

* Body weight 75-95kg, BMI 18.0-32.0 kg/m^2
* Refrain from sperm donation 110 days after dosing

Exclusion Criteria:

* Current or recent gastrointestinal disease
* Any GI surgery that could impact drug absorption
* Active, known, or suspected autoimmune disease

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male inclusion only
Enrollment: 9 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time Zero to Time of Last Quantifiable Concentration (AUC[0-T]) | up to 28 days
  Measured by plasma concentrations
Percent of Total Radioactivity Recovered in All Excreta (% total) | up to 28 days
  Measured by plasma urine, feces, and vomit (if applicable) volumes and radioactivity counts
Half-Life (T-HALF) | up to 28 days
  Measured by plasma concentrations
Total Body Clearance (CLT) | up to 28 days
  Measured by plasma concentrations
Volume of Distribution during Terminal Elimination Phase (Vz/F) | up to 28 days
  Measured by plasma concentrations
Time to Maximum Observed Concentration (Tmax) | up to 28 days
  Measured by plasma concentrations

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | up to 28 days
  Measured by investigator assessment
Results of electrocardiogram tests (ECGs) | up to 28 days
  Measured by investigator assessment
Results of vital sign measurements | up to 28 days
  Measured by investigator assessment
Results of clinical laboratory tests | up to 28 days
  Measured by investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol- Myers Squibb, Principal Investigator — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/